CLINICAL TRIAL: NCT01435382
Title: A Phase 1, Open-label, Randomized, Single Dose, Parallel Group Study To Assess The Pharmacokinetics And Pharmacodynamics Of Pf-04950615 Following Subcutaneous And Intravenous Doses In Adult Subjects With Hypercholesterolemia
Brief Title: A Pharmacokinetic and Pharmacodynamic Study of PF-04950615 (RN316) in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1481006
Record Dates: First submitted 2011-09-07; First posted 2011-09-16 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-10

CONDITIONS: Hypercholesterolemia; Dyslipidemias; Hyperlipidemias; Lipid Metabolism Disorders; Metabolic Diseases
Keywords: PF-04950615; RN316
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Hyperlipidemias; Lipid Metabolism Disorders; Metabolic Diseases | interventions — bococizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental)
  Interventions: Biological: PF-04950615 (RN316)
- Group B (Experimental)
  Interventions: Biological: PF-04950615 (RN316)
- Group C (Experimental)
  Interventions: Biological: PF-04950615 (RN316)
- Group D (Experimental)
  Interventions: Biological: PF-04950615 (RN316)

INTERVENTIONS:
Biological: PF-04950615 (RN316) — Dose A - single-dose intravenous infusion
  Arms: Group A
Biological: PF-04950615 (RN316) — Dose B - single-dose subcutaneous injection
  Arms: Group B
Biological: PF-04950615 (RN316) — Dose C - single-dose subcutaneous injection
  Arms: Group C
Biological: PF-04950615 (RN316) — Dose D - single-dose subcutaneous injection
  Arms: Group D

SUMMARY:
This Phase 1 study has been designed to evaluate the absolute bioavailability of PF-04950615 (RN316) in subjects with hypercholesterolemia who are not currently on lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C greater than or equal to 130 mg/dL at two qualifying screening visits.
* Total body weight greater than or equal to 50 kg (110 lbs) and less than or equal to 150 kg (330 lbs)

Exclusion Criteria:

* Lipid-lowering prescription medications, homeopaths, herbal medicines, or nutritional supplements.
* Poorly controlled type 1 or type 2 diabetes.
* History of a cardiovascular or cerebrovascular event or related procedure during the past year.
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Elite Research Institute, Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - PAREXEL International - Baltimore Early Phase Clinical Unit, Baltimore, Maryland
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Prism Research, Saint Paul, Minnesota
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Udata C, Garzone PD, Gumbiner B, Joh T, Liang H, Liao KH, Williams JH, Meng X. A Mechanism-Based Pharmacokinetic/Pharmacodynamic Model for Bococizumab, a Humanized Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, and Its Application in Early Clinical Development. J Clin Pharmacol. 2017 Jul;57(7):855-864. doi: 10.1002/jcph.867. Epub 2017 Feb 9. PMID 28181260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481006&StudyName=A%20Pharmacokinetic%20and%20Pharmacodynamic%20Study%20of%20PF-04950615%20%28RN316%29%20in%20Subjects%20with%20Hypercholesterolemia

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04950615 IV 200 mg: Participants received single intravenous (IV) infusion dose of PF-04950615 200 milligram (mg) on Day 1. Participants were followed up to Day 85.
- PF-04950615 SC 200 mg (2 Injections of 1 mL): Participants received subcutaneous (SC) dose of PF-04950615 200 mg on Day 1; 2 injections (100 milligram per milliliter [mg/mL]) of 1 milliliter (mL) each at two different quadrants of the abdomen; 1 injection per quadrant. Participants were followed up to Day 85.
- PF-04950615 SC 200 mg (1 Injection of 2 mL): Participants received single SC dose of PF-04950615 200 mg on Day 1; 1 injection (100 mg/mL) of 2 mL. Participants were followed up to Day 85.
- PF-04950615 SC 100 mg (1 Injection of 1 mL): Participants received single SC dose of PF-04950615 100 mg on Day 1; 1 injection (100 mg/mL) of 1 mL. Participants were followed up to Day 85.
Period: Overall Study
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Started | 12 | 13 | 13 | 11
Completed | 11 | 11 | 12 | 10
Not Completed | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL) | Total
Number analyzed (Participants) | 12 | 13 | 13 | 11 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.9) | 55.6 (9.8) | 52.1 (6.9) | 53.2 (12.3) | 52.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 6 | 21
  Male | 8 | 9 | 6 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04950615
Time Frame: Pre-dose, 30 minutes, 1, 8, 24, 48, 72, 96, 120, 168, 336, 504, 672, 840, 1008, 1176, 1344, 1512, 1680, 2016 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all participants randomized and treated who have at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
nanogram per milliliter (ng/mL) | 65810 (14047) | 15900 (18289) | 8922 (4016.4) | 10470 (18219)

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04950615
Time Frame: as for outcome 1
Population: PK parameter analysis population included all participants randomized and treated who have at least 1 of the PK parameters of primary interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
hour | 1.00 [1.00 to 1.08] | 95.2 [8.00 to 167] | 96.0 [71.0 to 167] | 72.0 [8.00 to 504]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of PF-04950615
Time Frame: as for outcome 1
Population: PK parameter analysis population included all participants randomized and treated who have at least 1 of the PK parameters of primary interest. Here 'N' (Overall Number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 11 | 13 | 13 | 11
nanogram*hour per milliliter | 13360000 (3635200) | 3420000 (2024100) | 2862000 (1638000) | 1529000 (849890)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero To Infinity (AUCinf) of PF-04950615
Time Frame: as for outcome 1
Population: PK parameter analysis population included all participants randomized and treated who have at least 1 of the PK parameters of primary interest. Here 'N' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 11 | 10 | 11 | 7
nanogram*hour per milliliter | 13510000 (3644400) | 3911000 (2008600) | 3173000 (1728000) | 1271000 (411160)

5. Primary Outcome: Apparent Clearance (CL/F) of PF-04950615 Subcutaneous Groups
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance (CL/F) is influenced by the fraction of the dose absorbed from plasma after SC administration of drug.
Time Frame: as for outcome 1
Population: PK parameter analysis population included all participants randomized and treated who have at least 1 of the PK parameters of primary interest. Here 'N' signifies those participants who were evaluable for this measure. This outcome measure was planned not to be analyzed in reporting arm: PF-04950615 IV 200 mg.
Measure: Mean (Standard Deviation); unit: milliliter per hour
Arm/Group | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 10 | 11 | 7
milliliter per hour | 71.64 (53.293) | 80.08 (42.654) | 85.54 (26.453)

6. Primary Outcome: Clearance (CL) of PF-04950615 Intravenous Group
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: PK parameter analysis population. Here 'N' signifies those participants who were evaluable for this measure. This outcome measure was planned not to be analyzed in reporting arms: PF-04950615 SC 200 mg (2 injections of 1mL), PF-04950615 SC 200 mg (1 injection of 2 mL) and PF-04950615 SC 100 mg (1 injection of 1 mL).
Measure: Mean (Standard Deviation); unit: milliliter per hour
Arm/Group | PF-04950615 IV 200 mg
Number analyzed (Participants) | 11
milliliter per hour | 15.82 (4.3037)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of PF-04950615 Subcutaneous Groups
Description: Volume of distribution (Vz) is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction of the dose absorbed from plasma after SC administration of drug.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 10 | 11 | 7
milliliter | 17770 (13555) | 19400 (19371) | 18400 (6381.5)

8. Primary Outcome: Volume of Distribution at Steady State (Vss) of PF-04950615 Intravenous Group
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is determined when overall intake of drug is in dynamic equilibrium with its elimination.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | PF-04950615 IV 200 mg
Number analyzed (Participants) | 11
milliliter | 4232 (757.77)

9. Primary Outcome: Terminal Elimination Half-life (t1/2) of PF-04950615
Description: t1/2 is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 11 | 10 | 11 | 7
hour | 202.4 (76.391) | 187.6 (87.298) | 153.2 (49.106) | 152.6 (43.324)

10. Primary Outcome: Absolute Bioavailability of PF-04950615 Subcutaneous Groups
Description: Bioavailability is defined as the rate and extent to which the active moiety administered drug reaches the systemic circulation. Absolute bioavailability of the subcutaneous doses was estimated by comparing log-transformed dose-normalized AUClast for subcutaneous to intravenous dose.
Time Frame: as for outcome 1
Population: PK parameter analysis population included all participants randomized and treated who have at least 1 of the PK parameters of primary interest. Here 'N' signifies those participants who were evaluable for this measure. This outcome measure was not analyzed in reporting arm: PF-04950615 IV 200 mg.
Measure: Number (95% Confidence Interval); unit: percentage of bioavailability
Arm/Group | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 13 | 13 | 11
percentage of bioavailability | 20.60 [13.74 to 30.87] | 21.24 [14.40 to 31.33] | 19.54 [13.25 to 28.83]

11. Secondary Outcome: Absolute Value of Fasting Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: Day 2, 3, 4, 5, 6, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85
Population: Pharmacodynamic (PD) population included all participants randomized and treated who had at least 1 plasma concentration of PF-04950615, and lipid panel or proprotein convertase subtilisin/kexin type 9 (PCSK9) data. Here, "Number of participants analyzed" signifies number of participants evaluable at different time points.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
milligram per deciliter (mg/dL)
  Day 2 | 154.00 (30.899) | 145.15 (29.653) | 148.31 (29.965) | 143.36 (24.250)
  Day 3 | 147.33 (23.274) | 132.54 (27.933) | 138.31 (26.961) | 134.18 (26.294)
  Day 4: number analyzed (Participants) | 11 | 13 | 13 | 11
  Day 4 | 131.09 (20.637) | 119.08 (31.481) | 125.77 (29.936) | 126.55 (27.883)
  Day 5 | 126.67 (26.476) | 104.46 (33.301) | 116.46 (38.937) | 119.91 (31.995)
  Day 6 | 128.92 (34.828) | 91.38 (26.355) | 101.31 (30.872) | 111.55 (29.733)
  Day 8: number analyzed (Participants) | 10 | 13 | 13 | 10
  Day 8 | 96.70 (17.257) | 91.92 (40.016) | 93.85 (32.695) | 104.20 (20.896)
  Day 15: number analyzed (Participants) | 11 | 12 | 12 | 11
  Day 15 | 68.73 (18.906) | 69.67 (25.115) | 69.83 (29.649) | 73.00 (26.069)
  Day 22: number analyzed (Participants) | 11 | 11 | 13 | 11
  Day 22 | 60.27 (14.143) | 82.45 (38.508) | 72.85 (28.801) | 103.18 (32.230)
  Day 29: number analyzed (Participants) | 11 | 11 | 12 | 11
  Day 29 | 65.82 (11.303) | 126.18 (45.683) | 115.75 (24.984) | 142.64 (23.243)
  Day 36: number analyzed (Participants) | 11 | 10 | 12 | 10
  Day 36 | 74.73 (23.749) | 125.10 (34.962) | 133.75 (24.458) | 140.80 (25.529)
  Day 43: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 43 | 96.00 (33.308) | 142.45 (33.255) | 140.75 (26.362) | 149.60 (27.261)
  Day 50: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 50 | 119.64 (28.790) | 149.45 (49.178) | 152.17 (25.074) | 151.70 (29.691)
  Day 57: number analyzed (Participants) | 10 | 11 | 12 | 10
  Day 57 | 150.20 (26.931) | 155.73 (35.755) | 152.25 (21.192) | 163.40 (38.839)
  Day 64: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 64 | 155.27 (36.072) | 154.09 (30.164) | 148.33 (20.637) | 152.00 (32.139)
  Day 71: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 71 | 151.00 (27.928) | 149.91 (32.473) | 148.00 (16.432) | 141.80 (26.561)
  Day 85: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 85 | 159.82 (21.577) | 151.00 (26.461) | 153.50 (28.688) | 137.30 (18.325)

12. Secondary Outcome: Percent Change From Baseline in Fasting Low-density Lipoprotein Cholesterol (LDL-C) at Day 2, 3, 4, 5, 6, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71 and 85
Description: Baseline was the average of observations collected on Days 7 and 1 prior to the study treatment administration.
Time Frame: Baseline, Day 2, 3, 4, 5, 6, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 85
Population: PD population included all participants randomized and treated who had at least 1 plasma concentration of PF-04950615, and lipid panel or PCSK9 data. Here, "Number of Participants Analyzed" signifies number of participants evaluable at different time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
percent change
  Day 2 | -5.93 (13.438) | -7.89 (11.329) | -7.05 (8.311) | -8.05 (10.310)
  Day 3 | -9.85 (7.085) | -16.31 (8.049) | -13.06 (9.137) | -14.27 (11.100)
  Day 4: number analyzed (Participants) | 11 | 13 | 13 | 11
  Day 4 | -17.87 (8.076) | -25.44 (9.346) | -21.20 (12.194) | -19.40 (11.037)
  Day 5 | -22.59 (11.972) | -34.84 (13.442) | -28.05 (16.909) | -23.83 (14.811)
  Day 6 | -21.59 (17.003) | -42.14 (12.827) | -36.62 (14.459) | -29.14 (13.507)
  Day 8: number analyzed (Participants) | 10 | 13 | 13 | 10
  Day 8 | -40.81 (13.225) | -43.18 (17.765) | -41.47 (16.099) | -34.00 (9.161)
  Day 15: number analyzed (Participants) | 11 | 12 | 12 | 11
  Day 15 | -58.13 (12.698) | -56.25 (13.925) | -56.45 (18.729) | -53.43 (14.985)
  Day 22: number analyzed (Participants) | 11 | 11 | 13 | 11
  Day 22 | -63.97 (7.455) | -48.49 (19.518) | -54.63 (15.528) | -34.63 (15.892)
  Day 29: number analyzed (Participants) | 11 | 11 | 12 | 11
  Day 29 | -60.61 (5.751) | -19.57 (23.437) | -27.49 (16.364) | -8.06 (14.174)
  Day 36: number analyzed (Participants) | 11 | 10 | 12 | 10
  Day 36 | -55.43 (13.394) | -20.45 (19.212) | -15.45 (20.597) | -9.42 (12.159)
  Day 43: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 43 | -42.94 (17.217) | -8.62 (14.204) | -10.12 (25.814) | -3.61 (13.949)
  Day 50: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 50 | -28.72 (14.755) | -5.91 (17.374) | -4.41 (15.372) | -2.38 (15.363)
  Day 57: number analyzed (Participants) | 10 | 11 | 12 | 10
  Day 57 | -10.00 (12.039) | -0.77 (10.237) | -4.63 (10.493) | 4.51 (17.233)
  Day 64: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 64 | -7.59 (15.843) | -1.17 (9.787) | -6.94 (11.837) | -1.90 (19.561)
  Day 71: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 71 | -9.93 (10.904) | -4.10 (11.984) | -6.95 (10.454) | -8.87 (11.161)
  Day 85: number analyzed (Participants) | 11 | 11 | 12 | 10
  Day 85 | -3.67 (14.381) | -2.21 (15.821) | -3.47 (18.833) | -10.76 (13.458)

13. Secondary Outcome: Duration of Fasting LDL-C Suppressed Below 70 mg/dL and 100 mg/dL
Time Frame: Day 1 up to Day 85
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
days
  Below 70 mg/dL: number analyzed (Participants) | 11 | 9 | 8 | 4
  Below 70 mg/dL | 9.4 (8.25) | 8.7 (7.55) | 7.5 (7.62) | 4.5 (4.04)
  Below 100 mg/dL: number analyzed (Participants) | 12 | 13 | 12 | 11
  Below 100 mg/dL | 21.8 (12.64) | 12.3 (10.43) | 12.8 (9.83) | 8.8 (8.10)

14. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state.
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
Participants
  Adverse Events | 7 | 7 | 8 | 6
  Serious Adverse Events | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Number of Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event) and severe (caused problem that interferes significantly with usual activities or the clinical status, study drug stopped due to adverse event).
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Number; unit: adverse events
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
adverse events
  Mild | 12 | 14 | 13 | 5
  Moderate | 0 | 2 | 6 | 2
  Severe | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Number of Participants With Treatment Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
Participants
  Adverse Events | 3 | 3 | 1 | 1
  Serious Adverse Events | 0 | 0 | 0 | 0

17. Other Pre Specified Outcome: Number of Participants With Injection Site Reactions
Description: The injection site reaction included erythema, induration, ecchymosis, injection site pain, injection site pruritus.
Time Frame: Day 1 up to Day 3
Population: Safety analysis set included all participants who had at least 1 dose of study medication. This outcome measure was planned not to be analyzed in reporting arm: PF-04950615 200 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 13 | 13 | 11
Participants | 2 | 5 | 4

18. Other Pre Specified Outcome: Number of Injection Site Reactions Reported as Adverse Events
Description: The injection site reactions included erythema, induration, ecchymosis, injection site pain and injection site pruritus. An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Day 1 up to Day 3
Population: Safety analysis set included all participants who had at least 1 dose of study medication. This outcome measure was planned not to be analyzed in reporting arm: PF-04950615 200 mg IV.
Measure: Number; unit: injection site reactions
Arm/Group | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 13 | 13 | 11
injection site reactions | 0 | 0 | 0

19. Other Pre Specified Outcome: Visual Analogue Scale (VAS)
Description: Participants indicated the amount of pain experienced due to study drug injection, on a VAS of 0 (no pain) to 100 (very severe pain), where higher scores indicate higher intensity of pain.
Time Frame: Day 1: Immediately post-dose, 0.5, 1.0, 2.0, 8.0 hours post-dose; Day 2, 3
Population: Safety analysis set included all participants who had at least 1 dose of study medication. Here, "Number of Participants Analyzed" signifies number of participants evaluable at different time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PF-04950615 SC 200 mg (2 Injections of 1mL): Injection 1: Participants received single SC dose of PF-04950615 200 mg on Day 1; 1 injection (100 mg/mL) of 1 mL at one quadrant of the two quadrants in abdomen. Participants were followed up to Day 85.
- PF-04950615 SC 200 mg (2 Injections of 1mL): Injection 2: Participants received single SC dose of PF-04950615 200 mg on Day 1; 1 injection (100 milligram per milliliter [mg/mL]) of 1 milliliter (mL) at second quadrant of the two quadrants in abdomen. Participants were followed up to Day 85.
Arm/Group | PF-04950615 SC 200 mg (2 Injections of 1mL): Injection 1 | PF-04950615 SC 200 mg (2 Injections of 1mL): Injection 2 | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 13 | 13 | 13 | 11
units on a scale
  Day 1: Immediately post-dose | 3.678 (4.8618) | 2.308 (2.3232) | 3.824 (7.7523) | 3.273 (3.3194)
  Day 1: 0.5 hour | 1.462 (1.4500) | 1.769 (1.8328) | 3.208 (7.0388) | 1.455 (2.2962)
  Day 1: 1.0 hour | 1.231 (1.3009) | 1.462 (1.4500) | 1.228 (1.8771) | 1.364 (1.4334)
  Day 1: 2.0 hours | 1.651 (1.5021) | 1.462 (1.5064) | 1.305 (1.8874) | 1.455 (2.0181)
  Day 1: 8.0 hours | 1.231 (1.4806) | 1.308 (1.3775) | 1.077 (1.7541) | 1.182 (1.5374)
  Day 2 | 1.077 (1.3205) | 1.461 (1.5610) | 1.230 (2.1663) | 1.364 (1.5015)
  Day 3: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 3 |  | 0.990 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. |  |

20. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory parameters evaluated for abnormalities were: hematology (hemoglobin [Hgb], hematocrit, red blood cell [RBC] count, platelets, white blood cell count [WBC], lymphocytes, total neutrophils, basophils, eosinophils, monocytes); coagulation (partial thromboplastin time, prothrombin time [PT], PT international ratio); clinical chemistry (glucose, creatine kinase, amylase, lipase); liver function (total, direct and indirect bilirubin, aspartate aminotransferase [AT], alanine AT, gamma-glutamyl transferase, alkaline phosphatase, total protein, albumin, lactate dehydrogenase); renal function (blood urea nitrogen, creatinine, uric acid); urinalysis (urine- specific gravity, pH, glucose, ketones, blood/Hgb, nitrite, leukocyte, esterase, RBC, WBC, epithelial cells, hyaline cast and bacteria); lipid (cholesterol); electrolytes (sodium, potassium, chloride, calcium, magnesium, phosphate, bicarbonate). Clinical significance of laboratory abnormalities were judged by investigator.
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- PF 04950615 SC 100 mg (1 Injection of 1 mL): Participants received single SC dose of PF-04950615 100 mg on Day 1; 1 injection (100 mg/mL) of 1 mL. Participants were followed up to Day 85.
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF 04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
Participants | 0 | 0 | 0 | 0

21. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs abnormalities included: maximum increase or decrease from baseline in supine systolic blood pressure (BP) greater than or equal to (>=) 30 millimeter of mercury (mmHg); maximum increase or decrease from baseline in supine diastolic BP of >=20 mmHg; supine pulse rate less than (<) 40 beats per minute (bpm) and greater than (>) 120 bpm; standing pulse rate less than (<) 40 beats per minute (bpm) and greater than (>) 140 bpm. Clinical significance of vital signs were judged by investigator.
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
Participants | 1 | 1 | 4 | 2

22. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG)
Description: ECG abnormalities included 1) PR interval: maximum >=300 maximum millisecond (msec), increase of >=25 percent (%) for baseline value of >200 msec and maximum increase of >=50% for baseline value of less than or equal to (<=) 200 msec; 2) QRS interval: maximum >=200 msec, maximum increase of >=25 % for baseline value of >100 msec and maximum increase of >=50% for baseline value of <=100 msec; 3) QT interval corrected using the Fridericia's formula (QTCF): 450 msec to <= 480 msec, 480 msec to <=500 msec, > 500 msec, maximum increase from baseline of >30 to <=60 msec and maximum increase from baseline of >60 msec. Clinical significance of ECG were judged by investigator.
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
Participants | 0 | 0 | 0 | 0

23. Other Pre Specified Outcome: Percentage of Participants With Positive Anti-drug (Anti-PF 04950615) Antibodies
Description: Human serum samples of participants who received PF-04950615 were analyzed for the presence of anti-PF-04950615 antibodies by using the semi quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1 up to Day 85
Population: Safety analysis set included all participants who had at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF 04950615 SC 100 mg (1 Injection of 1 mL)
Number analyzed (Participants) | 12 | 13 | 13 | 11
percentage of participants | 8.3 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04950615 IV 200 mg | PF-04950615 SC 200 mg (2 Injections of 1 mL) | PF-04950615 SC 200 mg (1 Injection of 2 mL) | PF-04950615 SC 100 mg (1 Injection of 1 mL)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 7/12 | 7/13 | 8/13 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04950615 IV 200 mg (N=12) | PF-04950615 SC 200 mg (2 Injections of 1 mL) (N=13) | PF-04950615 SC 200 mg (1 Injection of 2 mL) (N=13) | PF-04950615 SC 100 mg (1 Injection of 1 mL) (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crying (General disorders) | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 3 | 4
Viral infection (Infections and infestations) | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 3 | 1
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.